CLINICAL TRIAL: NCT04663451
Title: An Assessment of the Occurrence of Hypothyroidism in Patients Treated With RAI For Hyperthyroidism, And it's Prognostic Factors.
Brief Title: An Assessment of the Occurrence of Hypothyroidism in Patients Treated With RAI for Hyperthyroidism.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Brigitte Velkeniers, Head of the department of Internal Medicine and Endocrinology, Universitair Ziekenhuis Brussel
Other Study IDs: 2019/435
Record Dates: First submitted 2020-11-26; First posted 2020-12-11 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Nodule Solitary Thyroid; Toxic Multinodular Goiter; Radioactive Iodine-Induced Hypothyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Toxic Nodule: Hyperthyroid patients with underlying toxic nodule
  Interventions: Radiation: radioacive iodine therapy
- Toxic multinodular goiter: Hyperthyroid patients with underlying toxic multinodular goiter
  Interventions: Radiation: radioacive iodine therapy

INTERVENTIONS:
Radiation: radioacive iodine therapy — Hyperthyroid patients who have undergone radioactive iodine treatment to cure them from their hyperthyroidism.

SUMMARY:
Low RAIU in patients with hyperthyroidism represents a common obstacle in the treatment with RAI. Therefore, a higher dose of RAI must be administered to cure hyperthyroidism in these patients. If we treat patients with thiamazole before starting RAI treatment, serum TSH will rise and result in an increase in iodine uptake by the thyroid gland. By doing so, the dose of RAI to be administered might be lowered to achieve similar therapeutic efficacy.

In the past, either calculated or fixed doses of 131I have been used to treat hyperthyroidism. The supposed advantage of a calculated dose compared to a fixed dose is the lowering of hypothyroidism frequency. However, various research papers have contradicted this statement.

Antithyroid drugs and RAI therapy have been widely used in the past, either in combination, or independent from one another. This has been done primarily in older patients, to reduce the risk of exacerbation of hyperthyroid symptoms after initiation of RAI.

The use of propylthiouracil has been shown to decrease the response rate after RAI due to radioprotective effects.

The use of methimazole and carbimazole did not have a negative effect on treatment failure, as long as the medication was discontinued various days before RAI administration. Although this statement is contested in other studies.

It is interesting to evaluate retrospective data of patients treated with RAI to evaluate prognostic factors of treatment respons and post RAI hypothyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Hyperthyroid patients, either subclinical or overt, who have undergone RAI treatment in the period of 2005-2015.

Exclusion Criteria:

* Prior use of L-thyroxine
* Prior thyroid surgery
* Prior RAI treatment
* Patients with thyroiditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hyperthyroid patients, either subclinical or overt, who have undergone RAI treatment in the time period of 2005-2015. They have underlying toxic multinodular goiter or a toxic nodule.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients in which hypothyroidism occurs | Within 1 year after treatment
  The proportion of patients in which hypothyroidism occurs after radioiodine treatment
The proportion of patients in which hypothyroidism occurs | Between 1-2 years after treatment
  The proportion of patients in which hypothyroidism occurs after radioiodine treatment
The proportion of patients in which hypothyroidism occurs | Between 2-5 years after treatment
  The proportion of patients in which hypothyroidism occurs after radioiodine treatment

CONTACTS AND LOCATIONS:
Overall Officials: Corina Andreescu, Doctorate, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
The data may be shared with other researchers to continue this type of research in this particular domain and to answer further questions that arise from the process of this study.